CLINICAL TRIAL: NCT04744909
Title: Navigation System for Percutaneous Tracheotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Ullman, Associate professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SafeTrach 1
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Ventilation Therapy; Complications; Tracheostomy Complication
Keywords: Tracheotomy; tracheostomy; percutaneous dilatational tracheotomy; intensive care
MeSH Terms: interventions — Tracheotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous tracheotomy using a new device (Experimental)
  Interventions: Device: SafeTrach for tracheotomy

INTERVENTIONS:
Device: SafeTrach for tracheotomy — The navigation system is a forceps-like instrument with an outer and an inner shank. The inner shank serves as a ventilation lumen and stabilizes the orotracheal tube in the midline of trachea. The outer shank acts as a three-dimensional guide for the puncturing needle to the midline of trachea

SUMMARY:
We have studied a new technique for percutaneous tracheotomy. The instrument gives a three dimensional positioning of the puncture. The technique is used on patients on ENT surgery and intensiv care.

DETAILED DESCRIPTION:
Percutaneous tracheotomy is a well-established method. Anatomical landmarks need to be identified. We introduce a new method that increases precision through three-dimensional navigation with a new instrument - SafeTrach.

SafeTrach is a pliers-like instrument. The inner shank acts as a ventilation tube while stabilizing the orotracheal tube in the trachea. The outer shank acts as a three-dimensional control instrument for the puncture needle.

We determined the puncture level in 20 patients using SafeTrach. We found that the distance from the vocal cords to the puncture site was about 45 mm for men and 42 mm for women. This was based on intraoperative measurements. In 13 patients, we studied the distance between the vocal cords and the optimal puncture site between the 2nd and 3rd tracheal ring with CT and found that the mean distance for men was 49.8 mm and for women 42.2 mm. We have used internal measurements in another 12 patients as follows: The orotracheal tube is positioned so that the proximal part of the cuff is just below the vocal cords. 2. The position of the tube is measured against the front teeth. 3. The orotracheal tube together with the inner shank is pulled up about 15 mm for both men and women. This means that part of the cuff lies between the vocal cords and you get an acceptable placement of the puncture needle.

By using SafeTrach you can use internal landmarks to indicate the puncture level. The positioning of the leg is done with high precision because SafeTrach acts as a stable guide. The navigation system minimizes the risk of extubation and damage to the posterior tracheal wall.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years old
* Patients requiring PDT for prolonged mechanical ventilation, airway protection or weaning failure

Exclusion Criteria:

* Pediatric patients
* Emergency tracheotomies
* Anatomical abnormalities due to hematoma/tumor/scarring from previous neck surgery/thyromegaly/unstable C-spine and difficult local anatomy. (Patients with obesity are not considered to be a hindrance for the SafeTrach technique as the location for puncture easily can be decided with help of the outer and inner shanks).
* Contra indication for re-intubation (suspected loss of airway during re-intubation)
* Coagulation abnormalities - INR>1.5, PTT >40, thrombocyte count <50.000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Navigation System for Percutaneous Tracheotomy | 30 minutes
  Precision of puncture site

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Karling, Ph.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden